CLINICAL TRIAL: NCT03491995
Title: A Unique Quadruple Regimen for of Helicobacter Pylori
Brief Title: A Unique Regimen for Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Helicobacter study
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadruple therapy (Experimental): Moxifloxacin, Nitazoxanide, Omeprazole sodium bicarbonate, Doxycyclin
  Interventions: Drug: Quadruple therapy
- Classic treatment (Active Comparator): Omeprazole, clarithromycin, amoxicillin
  Interventions: Drug: Classic treatment

INTERVENTIONS:
Drug: Quadruple therapy — Moxifloxacin, omeprazole sodium bicarbonate, nitazoxanide, doxycyclin
  Other Names: Moxiflox, Downoprazol, Nanazoxid, Doxymycin
  Arms: Quadruple therapy
Drug: Classic treatment — Omeprazole, amoxycillin, clarithromycin
  Other Names: Downoprazol, Emox, Klacid
  Arms: Classic treatment

SUMMARY:
The triple treatment including Proton pump inhibitor (PPI) -clarithromycin and amoxicillin or metronidazole was proposed 30 years ago at the first Maastricht conference to treat helicobacter pylori (H. pylori) infection and since that time, it has become the universal and standard treatment for helicobacter pylori.

However, the efficacy of this triple regimen has been seriously challenged, and they are gradually becoming ineffective

DETAILED DESCRIPTION:
Growing rates of treatment failure are observed worldwide and the eradication rate of triple therapy has declined over the past few decades. Helicobacter pylori infection has become increasingly resistant to traditional first line treatment regimens because of emerging antibiotic resistance coupled with poor patient compliance with completing the treatment course that decrease H. pylori eradication rates .So there is a considerable interest in evaluating new antibiotic combinations and regimens .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged older than 21 years Presenting by Dyspepsia Infected by H. pylori (as proved by positive stool antigen test) Agreed to participate in the study and signed the consent

Exclusion Criteria:

* Patients who have received treatment with proton pump inhibitors within 2 weeks, NSAID or antibiotics within 4 weeks before study entry Patients who had received H pylori treatment before. Patients presenting by upper gastrointestinal bleeding Pregnant females Patients who have significant gastrointestinal, renal, hepatic, cardiovascular, metabolic, hematological disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with eradicated Helicobacter infection | 6 months
  Number of patients with eradicated infection

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Yousry, Prof, Principal Investigator — Head of Hepatology and infectious diseases dept.-Cairo University; Walied El-Hossary, MD, Study Director — Hepatology and infectious diseases dept.-Cairo University; Mohamed Alboraie, MD, Study Chair — Internal Medicine dept.-Alazhar University; Sherief Abd-Elsalam, MD, Study Chair — Hepatology and Infectious diseases- Tanta University; Asem Elfert, Prof, Study Chair — Hepatology and Infectious diseases- Tanta University; Hussein A Elamin, Prof, Study Chair — Internal Medicine-Assuit University; Mohamed Adel Elbasiony, MD, Study Chair — Internal Medicine- Mansoura University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided